CLINICAL TRIAL: NCT01607645
Title: Phase II Trial Examining Epigenetic Priming With Decitabine Followed by Idarubicin and Cytarabine for Patients With Relapsed or Refractory AML.
Brief Title: Decitabine Followed by Idarubicin and Cytarabine in Treating Patients With Relapsed or Refractory AML and MDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early because there were other competing protocols.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Derek Stirewalt, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2588.00; NCI-2012-00769 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Decitabine; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm1: decitabine, idarubicin, cytarabine (Experimental): Patients receive decitabine IV over 1 hour on days -4 to 0, cytarabine IV continuously over 24 hours on days 1-7, and idarubicin IV over 10-15 minutes on days 1-3.
  Interventions: Drug: decitabine; Drug: idarubicin; Drug: cytarabine
- Arm2: decitabine, idarubicin, cytarabine (Experimental): Patients receive decitabine IV over 1 hour on days -9 to -5 and cytarabine and idarubicin as in Arm I.
  Interventions: Drug: decitabine; Drug: idarubicin; Drug: cytarabine

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside

SUMMARY:
The goals of this study are to learn about the effectiveness, the side-effects, if waiting to give the idarubicin and cytarabine may change the side effects or effectiveness, and to identify factors to predict for responses to this therapy. The trial will examine combination of three chemotherapy drugs. These drugs are decitabine, idarubicin, and cytarabine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the morphologic complete remission (CR) rates using a decitabine (DAC)-priming followed by idarubicin (IDA) and cytarabine (ARAC) in patients with relapsed or refractory acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. To determine CR without minimal residual disease (CRMRD-), CR with incomplete blood count recovery (CRi), CR with minimal residual disease (CRMRD+), and CR with incomplete blood count recovery and with minimal residual disease (CRiMRD+) rates.

II. To estimate the frequency and severity of regimen-related toxicities.

III. To identify biomarkers (e.g., deoxyribonucleic acid [DNA] methylation and expression changes including interferon regulatory factor [IRF]8) associated with clinical responses.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive decitabine intravenously (IV) over 1 hour on days -4 to 0, cytarabine IV continuously over 24 hours on days 1-7, and idarubicin IV over 10-15 minutes on days 1-3.

ARM II: Patients receive decitabine IV over 1 hour on days -9 to -5 and cytarabine and idarubicin as in Arm I.

In both arms, treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* All patients except those with acute promyelocytic leukemia (APL) who have morphological diagnosis of myelodysplastic syndromes (MDS) refractory anemia with excess blasts (RAEB)-II or AML by World Health Organization (WHO) diagnostic criteria and have either refractory or early relapsed disease; NOTE:

  * Diagnosis of refractory or relapsed disease must be based on evaluation of a bone marrow (BM) aspirate or peripheral blood (PB) flow cytometry; other standard MDS and AML prognostic studies such as cytogenetics, flow, and molecular testing are highly recommended prior to initiating DAC
  * A previous BM evaluation or PB flow cytometry from an outside facility are acceptable if the results have been deemed to be adequate for confirming the diagnosis and staging by University of Washington (UW)/Seattle Cancer Care Alliance (SSCA)/Fred Hutchinson Cancer Research Center (FHCRC) review
  * A BM biopsy is not routinely required but should be obtained if the previous evaluation is not deemed to be adequate for confirming diagnosis and staging by UW/SCCA/FHCRC review
* Must have received at least one previous cycle of treatment for myelodysplastic syndrome (MDS) or AML and be either refractory as defined as not responded to this therapy or in early relapse as defined as developing recurrence of the disease within 12 months of obtaining a CR
* May have previously received demethylating agents (e.g., DAC, 5-azacytidine [5AZA]) or histone deacetylases (e.g., suberoylanilide hydroxamic acid) for their MDS or AML if these demethylating agents were not used in combination with systemic anthracycline and ARAC chemotherapy
* May have received hematopoietic growth factors, thalidomide/lenalidomide, signal transduction inhibitors, or low dose cytarabine (=< 20 mg/m2/day)
* May not have received any therapy for their MDS or AML other than hydroxyurea or leukapheresis for at least 14 days prior to start of the first dose of DAC; all non-hematologic toxicities must have resolved to < grade 2
* Must have a "simplified" treatment-related mortality (TRM) score =< 9.2
* Females of childbearing potential must have a negative pregnancy test prior to initiation of the protocol therapy; females are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 12 weeks after treatment discontinuation
* Patients with an active or history of other malignancies are eligible, if their projected overall survival for that malignancy is at least 6 months
* Prior hormonal therapy such as aromatase inhibitors, selective estrogen receptor modulators, estrogen receptor down-regulators, luteinizing hormone-releasing hormone (LHRH) agonists and antagonists, and anti-androgens, must be completed at least 30 days prior to initiation of protocol therapy and must remain off hormonal therapy until the patient has finished chemotherapy for their MDS-RAEBII or AML
* Direct bilirubin =< 2.5 mg/dL (assessed within 14 days prior to registration) unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis
* No known hypersensitivity to decitabine (DAC), aracytidine triphosphate (ARAC), or idarubicin hydrochloride (IDA)
* No clinical evidence of central nervous system (CNS) involvement with leukemia, unless a lumbar puncture confirms the absence of leukemic blasts in the cerebrospinal fluid (CSF)
* No prior positive test for the human immunodeficiency virus (HIV)
* No uncontrolled systemic infection

Exclusion Criteria:

* Previous therapy with demethylating agents (e.g., DAC, 5AZA, etc.) or histone deacetylases (e.g., suberoylanilide hydroxamic acid, etc.) that was combined with daunorubicin (DNR) or IDA and ARAC
* Patients with acute promyelocytic leukemia (APL)
* Known hypersensitivity to DAC, ARAC, or IDA
* Clinical evidence of CNS involvement with leukemia, unless a lumbar puncture confirms the absence of leukemic blasts in the CSF
* Prior positive test for HIV
* Uncontrolled systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* A "simplified" TRM score > 9.2
* Bilirubin > 2.5 mg/dl (assessed within 14 days prior to registration), unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis
* Patients who have a projected overall survival < 6 months due to malignancies other than MDS or AML
* Documented symptomatic congestive heart failure or a documented left ventricular ejection fraction < 40% assessed by multigated acquisition (MUGA), echocardiography, or heart catheterization within 21 days prior to start of decitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Stirewalt, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant were enrolled between 8/23/12 and 5/16/13 at the FHCRC
Groups:
- Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine): Patients receive decitabine IV over 1 hour on days -4 to 0, cytarabine IV continuously over 24 hours on days 1-7, and idarubicin IV over 10-15 minutes on days 1-3.
  decitabine: Given IV
  idarubicin: Given IV
  cytarabine: Given IV
- Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine): Patients receive decitabine IV over 1 hour on days -9 to -5 and cytarabine and idarubicin as in Arm I.
  decitabine: Given IV
  idarubicin: Given IV
  cytarabine: Given IV
Period: Overall Study
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine) | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.75 (16.46) | 34.67 (13.01) | 43.86 (16.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Morphologic CR
Description: Morphologic complete remission (CR): Absolute Neutrophil Count (ANC)≥1,000/uL, platelet count ≥100,000/uL, <5% Bone Marrow (BM) blasts, no Auer rods (cytoplasmic inclusions which result from an abnormal fusion of the primary (azurophilic) granules), no morphologic dysplasia, and no evidence of extramedullary disease
Time Frame: Participants were monitored up until the point when they went off study following completion of the treatment (3 months)
Measure: Number; unit: participants
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 4 | 3
participants
  CR | 2 | 0
  CRi-MRD (Minimal Residual Disease) | 1 | 0
  Refractory | 1 | 3

2. Secondary Outcome: Resistant Disease Defined as Patient Survives at Least 14 Days After Completion of the Last Dose of Induction or Re-induction But Has Persistent Leukemia in Peripheral Blood (PB) or BM
Time Frame: Assessed for up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 4 | 3
Participants | 1 | 3

3. Secondary Outcome: Cytogenetic Response Defined as no Detectable Cytogenetic Abnormality in a Subsequent BM Specimen After Induction or Re-induction
Time Frame: Assessed for up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 4 | 3
Participants | 3 | 0

4. Secondary Outcome: CRMRD- Defined as Morphologic CR Without Evidence of Minimal Residual Disease by Flow Cytometry, Cytogenetics, or Other Known Molecular Biomarkers
Time Frame: Assessed for up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 4 | 3
Participants | 2 | 0

5. Secondary Outcome: CRi Defined as Meeting All Criteria for a Morphologic CR But ANC Remains Less Than 1,000/μL and/or Platelet Count Less Than 100,000/μL
Time Frame: Assessed for up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

6. Secondary Outcome: CRMRD+ Defined as a Morphologic CR But With Minimal Residual Disease by Flow Cytometry, Cytogenetics, or Other Known Molecular Biomarkers
Time Frame: Assessed for up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

7. Secondary Outcome: CRiMRD+ Defined as Meeting All Criteria for a CRi But With Evidence of Minimal Residual Disease by Flow Cytometry, Cytogenetics, or Other Known Molecular Biomarkers
Time Frame: Assessed for up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 4 | 3
Participants | 1 | 0

8. Secondary Outcome: TRM With Each Course of Decitabine-priming, Idarubicin, and Cytarabine
Time Frame: Assessed for up to Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

9. Secondary Outcome: Frequency and Severity of Grade 3, 4, and 5 Toxicities With Each Course of Decitabine-priming, Idarubicin, and Cytarabine According to NCI Common Terminology Criteria for Adverse Events Version (CTCAE) 4.0
Time Frame: Assessed for up to 3 months after completion study treatment
Population: We have analyzed 4 and 3 patients in each arm, respectively. One patient in each of the arms completed 2 cycles of therapy. The numbers provided in the Outcome Measure Data Table in Frequency and Severity of Grade 3, 4, and 5 Toxicities are the numbers of patients with each specified event.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 4 | 3
Participants
  CYCLE 1 : Infection Grade 3 | 2 | 0
  CYCLE 1 : Infection Grade 4 | 0 | 1
  CYCLE 1 : Hepatobiliary Grade 3 | 0 | 1
  CYCLE 1 : Blood and Lymphatic Grade 3 | 3 | 1
  CYCLE 1 : Gastrointenstinal Grade 3 | 0 | 0
  CYCLE 2 : Infection Grade 3: number analyzed (Participants) | 1 | 1
  CYCLE 2 : Infection Grade 3 | 0 | 0
  CYCLE 2 : Infection Grade 4 | 0 | 0
  CYCLE 2 : Hepatobiliary Grade 3 | 0 | 0
  CYCLE 2 : Blood and Lymphatic Grade 3 | 1 | 0
  CYCLE 2 : Gastrointenstinal Grade 3 | 1 | 0

10. Secondary Outcome: Severe Prolonged Aplasia
Time Frame: Assessed for up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

11. Secondary Outcome: Duration of Severe Neutropenia Defined as an ANC Less Than 500
Time Frame: Assessed for up to 5 years
Population: No member of Arm II was eligible for evaluation for this Outcome Measure. Therefore, no data was collected for Arm II.
Measure: Mean (Full Range); unit: days
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 3 | 0
days | 65 [25 to 106] |

12. Secondary Outcome: Duration of Moderate Neutropenia Defined as an ANC Less Than 1000
Time Frame: Assessed for up to 5 years
Population: No member of Arm II was eligible for evaluation for this Outcome Measure. Therefore, no data was collected for Arm II.
Measure: Mean (Full Range); unit: days
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 3 | 0
days | 67 [30 to 106] |

13. Secondary Outcome: Duration of Thrombocytopenia Defined as Platelet Count Less Than 100,000
Time Frame: Assessed for up to 5 years
Population: No member of Arm II was eligible for evaluation for this Outcome Measure. Therefore, no data was collected for Arm II.
Measure: Mean (Full Range); unit: days
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Number analyzed (Participants) | 3 | 0
days | 51 [18 to 103] |

ADVERSE EVENTS:
Time Frame: The Adverse Events were assessed while the participants were receiving study specific treatment for up to 3 months after the start of the treatment.
Arm/Group | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine)
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/3
Other Adverse Events (participants affected / at risk) | 4/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) (N=4) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine) (N=3)
Grade 4 Infection (Infections and infestations) | 0 (0) | 1 (1) — Patient became septic with coag negative Staphylococcus, requiring prolonged hospitalization and IV antibiotics with blood pressure support
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Decitabine Day -4 to Day 0), Idarubicin, Cytarabine) (N=4) | Arm II (Decitabine (Day -9 to Day -5), Idarubicin, Cytarabine) (N=3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) — Expected Grade 3 febrile neutropenia
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2 abdominal pain
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) — Grade 1 hemorrhoids
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2 diarrhea
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 2 (2) — One patient with Grade 1; one patient with Grade 2; one patient with Grade 3
Infection (Infections and infestations) | 2 (5) | 0 (0) — 2 patients with grade 3 C. difficle; 1 patient with Grade 3 UTI; 1 patient with Grade 3 device related infection; 1 patient with Grade 3 lung infection
Joint pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Patient developed both, Grade 2 elbow and knee pain
Back Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Patient developed Grade 1 back pain
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) — One patient developed Grade 2 menorrhagia
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) — One patient developed Grade 2 thrombotic event

LIMITATIONS AND CAVEATS:
Early termination due to similar competing protocol, which made statistical evaluation of primary endpoint and any meaningful evaluation of secondary time points not feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No